CLINICAL TRIAL: NCT00672399
Title: A Placebo- and Positive-Controlled Study of the Electrophysiological Effects of a Single 10 μg Dose of Exenatide on the 12-Lead Electrocardiogram QT Interval in Healthy Subjects
Brief Title: Electrophysiological Effects of a Single 10 μg Dose of Exenatide on the 12-Lead Electrocardiogram QT Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H8O-EW-GWCI
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Subjects
Keywords: Amylin; Eli Lilly; exenatide; moxifloxacin
MeSH Terms: interventions — Exenatide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Period 1 = placebo exenatide/placebo moxifloxacin; Period II = exenatide/placebo moxifloxacin; Period III = placebo exenatide/moxifloxacin
  Interventions: Drug: exenatide; Drug: Moxifloxacin; Drug: Placebo
- Sequence 2 (Experimental): Period I = exenatide/placebo moxifloxacin; Period II = placebo exenatide/moxifloxacin; Period III = placebo exenatide/placebo moxifloxacin
  Interventions: Drug: exenatide; Drug: Moxifloxacin; Drug: Placebo
- Sequence 3 (Experimental): Period 1 = placebo exenatide/moxifloxacin; Period II = placebo exenatide/moxifloxacin; Period III = exenatide/placebo moxifloxacin
  Interventions: Drug: exenatide; Drug: Moxifloxacin; Drug: Placebo
- Sequence 4 (Experimental): Period I = placebo exenatide/moxifloxacin; Period II = exenatide/placebo moxifloxacin; Period III = placebo exenatide/placebo moxifloxacin
  Interventions: Drug: exenatide; Drug: Moxifloxacin; Drug: Placebo
- Sequence 5 (Experimental): Period I = placebo exenatide/placebo moxifloxacin; Period II = placebo exenatide/moxifloxacin; Period III = exenatide/moxifloxacin
  Interventions: Drug: exenatide; Drug: Moxifloxacin; Drug: Placebo
- Sequence 6 (Experimental): Period I = exenatide/placebo moxifloxacin; Period II = placebo exenatide/placebo moxifloxacin; Period III = placebo exenatide/moxifloxacin
  Interventions: Drug: exenatide; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: exenatide — Subcutaneously injected, 10 mcg, single doses
  Other Names: Byetta
Drug: Moxifloxacin — oral, 400 mg tablet, single doses
Drug: Placebo — Subcutaneously injucted in an amount equivalent to exenatide; or orally as a tablet identical in appearance to Moxifloxacin. Both are single doses

SUMMARY:
This Phase 1, randomized, three period, placebo- and positive-controlled,double-blind, double-dummy, crossover study will be performed with approximately 80 healthy male and female subjects. The effects of single doses of exenatide (10 μg, subcutaneous), moxifloxacin (400 mg, oral) or placebo(subcutaneous or oral) on QT interval will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18 and 65 years, inclusive.
* Have body mass index (BMI) between 19 and 35 kg/m2, inclusive.
* If females, are not of child-bearing potential due to surgical sterilisation (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Women with an intact uterus are deemed postmenopausal if they have had cessation of menses for at least 1 year or 6 to 12 months of spontaneous amenorrhea with follicle stimulating hormone >40 IU/mL; age ≥45 years; not taking oral contraceptives for at least 1 year; and otherwise healthy.
* Subjects receiving hormone replacement therapy (HRT) or thyroxine as replacement therapy may participate providing they have been on stable therapy for at least 3 months and have a normal thyroid stimulating hormone (TSH) value.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Known allergies to exenatide or excipients, moxifloxacin or related compounds, or a history of multiple adverse drug allergies of any origin.
* Family history of sudden death.
* Personal history of unexplained syncope within last year.
* History or presence of cardiovascular (myocardial infarction, cerebrovascular accident, venous thromboembolism), respiratory, hepatic, renal, GI, endocrine, haematological, or neurological disorders.
* Evidence or history of Long QT Syndrome or significant active cardiac disease (e.g., arrhythmia, hypertension, congestive heart failure, hypokalaemia, mitral valve regurgitation, endocarditis, coronary artery heart disease), or symptoms of angina pectoris or transient ischaemic attacks within the previous 6 months.
* Females who are lactating.
* Have previously completed or withdrawn from this study or any other study investigating exenatide.
* Evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Evidence of hepatitis C and/or positive hepatitis C antibody.
* Evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Use of over-the-counter or prescription medication (other than, for example, thyroid replacement, occasional intake of paracetamol, or vitamin or mineral supplements) 7 and 14 days, respectively, before dosing and throughout the study.
* Cumulative blood donation of more than 500 mL within the last 3 months.
* Subjects who have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or subjects unwilling to stop alcohol consumption for the duration of the study(1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Subjects who smoke or have smoked within 28 days of their screening visit and who are unable to abide by the study restrictions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Comparison of exenatide's effect on QT interval when compared to placebo | single doses - measurements at 1, 2, 3, 4, 5.5 and 10 hours after dosing
  To determine, in healthy subjects, that a single 10 μg dose of exenatide does not differ from placebo in the mean change from predose in 12-lead ECG correct QT (QTc) interval measurements

SECONDARY OUTCOMES:
Measurement of any QTcF changes following exenatide versus glucose, potassium, and insulin | single doses - samples drawn at and EKGs at -15 min, hours 1, 2, 3, 4, 5.5, 10
  To explore the influence of potential physiological covariates such as plasma insulin, plasma glucose, and potassium on QTc interval in healthy subjects
Assessment of plasma exenatide concentrations and QTc interval | During Periods I, II, and III, ECGs should be recorded at the following
  Evaluation of the relationship between plasma exenatide concentrations and QTc interval in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (2):
- United Kingdom (2):
  - Reseach Site, Derriford, Plymouth
  - Research Site, Leeds, West Yorkshire